CLINICAL TRIAL: NCT05341167
Title: Use of the Hypotension Prediction Index Algorithm (HPI) for the Prevention of Intraoperative Hypotension (IOH) in Adult Patients Undergoing Spinal Surgery: Study Protocol for a Randomized Clinical Trial
Brief Title: HPI Algorithm for the Prevention of IOH During Spinal Surgery [HPIFPIOH]
Acronym: HPIFPIOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Prof of Anestehsiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HPIFPIOH
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Hypotension
MeSH Terms: interventions — Vasoconstrictor Agents; Norepinephrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Double-Blinded clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Not aware of the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: (Active Comparator): The HPI algorithm will be used in order to prevent hypotensive episodes. When the HPI is greater than 85%, the anesthesiologist will have to intervene within the next 2 minutes taking the hemodynamic parameters available into consideration, as well as the treatment protocol that has been designed according to current literature
  Interventions: Device: HPI algorithm using Edwards device https://www.edwards.com/gb/devices/decision-software/hpi; Drug: Vasoactive Agent
- Control group: (Other): Hypotensive episodes will be treated with vasoactive agents and fluids according to the standard clinical practice. The HPI algorithm recordings will be blinded and will not be available to the anesthesiologist for the duration of the operation.
  Interventions: Drug: Vasoactive Agent

INTERVENTIONS:
Device: HPI algorithm using Edwards device https://www.edwards.com/gb/devices/decision-software/hpi — The HPI algorithm will be used in order to prevent hypotensive episodes. When the HPI is greater than 85%, the anesthesiologist will have to intervene within the next 2 minutes taking the hemodynamic parameters available into consideration, as well as the treatment protocol that has been designed according to current literature
  Other Names: noradrenaline; phenylephrine
  Arms: Intervention group:
Drug: Vasoactive Agent — Hypotensive episodes will be treated with vasoactive agents and fluids. The HPI algorithm recordings will be blinded and will not be available to the anesthesiologist for the duration of the operation.
  Other Names: noradrenaline; phenylephrine

SUMMARY:
The aim of this study is to investigate the hypothesis that the use of the Hypotension Prediction Index algorithm (HPI) can reduce intraoperative hypotension (IOH) in adult patients undergoing spinal surgery in the prone position under general anesthesia, as well as to explore its effect on in-hospital postoperative morbidity and mortality.

DETAILED DESCRIPTION:
The study is a Prospective Randomized clinical trial. Adult patients (>18y) undergoing spinal surgery in the prone position under general anesthesia will be included.

The patients will be randomized using a computer-generated, permuted block randomization with a 1:1 allocation into two groups.

Intervention group: in this group, the HPI algorithm will be used in order to prevent hypotensive episodes Control group: in this group standard anesthetic care will be provided. Hypotensive episodes will be treated with vasoactive agents and fluids.

All patients will receive the same type of anaesthesia (TIVA with propofol) and monitoring including Patient State Index (PSI), non-invasive monitoring of blood pressure, SpO2, continuous electrocardiographic monitoring, ETCO2 and urinary output. Additionally, invasive continuous measurement of the patient's blood pressure will be available via radial artery catheterization. The arterial catheter will be connected to both the standard monitor and the platform which includes the HPI software. Arterial blood gas testing will be performed on an hourly basis.

Intraoperative recordings include PSI values, hemodynamic parameters every 10-15 minutes and urinary output every hour. Hemodynamic parameters will also be collected electronically from the monitor. The total doses of propofol, opioids/sedatives, fluids and vasoactive agents will also be recorded, as well as the estimated blood loss.

In this study, time-weighted average (TWA) in hypotension will be calculated in all patients.[TWA= depth of hypotension x time spent in hypotension / total surgery time].

Postoperatively Blood sampling for hs-TropI will be collected after the surgical procedure and during the following 3 postoperative days. If an increase in the levels hs-Trop I is noted the patient will be inquired for symptoms of myocardial ischemia and a new ECG will be performed. A cardiology consultation will be requested, if necessary.

Creatinine levels and urinary output will be monitored during the first 2 postoperative days. Acute kidney injury will be assessed according to the AKIN classification.

All in-hospital incidents and in-hospital mortality will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing scheduled spine surgery performed in prone position under general anaesthesia

Exclusion Criteria:

* Heart failure with reduced ejection fraction (LVEF<35%)
* Severe aortic and/or mitral regurgitation
* Persistent atrial fibrillation or other significant cardiac arrhythmias
* Significant preoperative hypotension
* End-stage renal disease on dialysis/RRT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Time-weighted average (TWA) in hypotension | Up to 15 minutes after the end of operation
  Time-weighted average (TWA) in hypotension will be calculated in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Matsota, Prof, Principal Investigator — 2nd Department of Anesthesiology, Attikon University Hospital
Locations (2):
- Greece (2):
  - General Hospital of Athens "Georgios Gennimatas", Athens, Attica
  - Attikon Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilakouta Depaskouale MA, Archonta SA, Moutafidou SKappa, Paidakakos NA, Dimakopoulou AN, Matsota PK. Effectiveness of hypotension prediction index software in reducing intraoperative hypotension in prolonged prone-position spine surgery: a single-center clinical trial. J Clin Monit Comput. 2025 Oct;39(5):875-887. doi: 10.1007/s10877-025-01303-0. Epub 2025 May 23. PMID 40410627